CLINICAL TRIAL: NCT02672111
Title: An Open-Label Multicenter Study Assessing the Long-Term Safety of a Once-Weekly and Once-Monthly, Long-Acting Subcutaneous Injection Depot of Buprenorphine (CAM2038) in Adult Outpatients With Opioid Use Disorder
Brief Title: Long-Term Safety Study of Buprenorphine (CAM2038) in Adult Outpatients With Opioid Use Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braeburn Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-14-499
Record Dates: First submitted 2016-01-15; First posted 2016-02-03 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2019-07

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAM2038 q1w or q4w exposure to SL BPN/NX (Experimental): CAM2038 (buprenorphine FluidCrystal®)
  Subjects previously exposed to SL BPN/NX who received CAM2038 q1w or q4w
  Interventions: Drug: CAM2038 q1w or q4w exposure to SL BPN/NX
- CAM2038 q1w or q4w new to BPN treatment (Experimental): CAM2038 (buprenorphine FluidCrystal®) New to BPN Treatment who received CAM2038r q1w or q4w
  Interventions: Drug: CAM2038 q1w or q4w new to BPN treatment

INTERVENTIONS:
Drug: CAM2038 q1w or q4w exposure to SL BPN/NX
  Other Names: Buprenorphine injection
  Arms: CAM2038 q1w or q4w exposure to SL BPN/NX
Drug: CAM2038 q1w or q4w new to BPN treatment
  Other Names: Buprenorphine injection
  Arms: CAM2038 q1w or q4w new to BPN treatment

SUMMARY:
Open-label multi-center, 48 week safety study, consistent with standard practice for long-term safety studies. This one year safety study will utilize CAM2038 q1w (once weekly) and q4w (once monthly) and will have 3 phases: Screening, Treatment, and Follow-up.

DETAILED DESCRIPTION:
Open-label multi-center, 48 week safety study, consistent with standard practice for long-term safety studies. This one year safety study will utilize CAM2038 q1w (once weekly) and q4w (once monthly) and will have 3 phases: Screening, Treatment, and Follow-up.

Patients who are currently taking sublingual (SL) BPN (weekly or monthly prescription visits) or individuals who are actively seeking BPN treatment but who have not yet begun a treatment regimen, may be eligible for the study.

Following Screening, qualified subjects meeting inclusion criteria and not meeting exclusion criteria will be initiated on either CAM2038 q1w or q4w, based on their current treatment status (qualified subjects currently on SL BPN or seeking BPN treatment). Qualified subjects will be initiated or transitioned to CAM2038 q1w or q4w as follows:

Initiation of BPN treatment - initiate with CAM2038 q1w

Currently receiving SL BPN treatments - transfer to corresponding CAM2038 q1w or q4w dose

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to the conduct of any study-related procedures.
2. Male or female, 18-65 years of age, inclusive.
3. Female subjects of childbearing potential must be willing to use a highly effective method of contraception during the entire study (Screening Visit to Follow-Up Visit).
4. Current diagnosis of moderate or severe opioid use disorder (DSM-V) or past medical history of opioid use disorder currently being treated with SL BPN.
5. Considered by the Investigator to be a good candidate for BPN treatment, based on medical and psychosocial history.
6. Subjects must meet one of the following criteria for BPN treatment history:

   * Voluntarily seeking treatment for opioid use disorder (not currently on BPN treatment for at least last 60 days but seeking BPN treatment), or;
   * Currently on SL BPN treatment.

Exclusion Criteria:

1. Current diagnosis of Acquired Immune Deficiency Syndrome (AIDS).
2. Current diagnosis of chronic pain requiring opioids for treatment.
3. Current DSM-V diagnosis for moderate to severe substance use disorder (including alcohol) other than opioids, caffeine or nicotine and currently being treated as the primary substance use disorder.
4. Recent history of or current evidence of suicidal ideation or active suicidal behavior as based on the Columbia Suicide Severity Rating Scale (C-SSRS) ("Yes" responses to questions 4 or 5).
5. Pregnant or lactating or planning to become pregnant during the study.
6. Hypersensitivity or allergy to naloxone (only for subjects receiving the SL BPX test dose), BPN or excipients of CAM2038.
7. Requires chronic use of agents that are strong inhibitors or inducers of cytochrome P450 3A4 (CYP 3A4) such as some azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., clarithromycin), or protease inhibitors (e.g., ritonavir, indinavir, and saquinavir).
8. Hepatitis, unless under stable treatment, at the discretion of the Investigator.
9. Any pending legal action that could prohibit participation or compliance in the study.
10. Exposure to any investigational drug within the 4 weeks prior to Screening.
11. Aspartate aminotransferase (AST) levels ≥3 X the upper limit of normal, alanine aminotransferase (ALT), levels ≥ 3 X the upper limit of normal, total bilirubin ≥ 1.5 X the upper limit of normal, or creatinine ≥ 1.5 X upper limit of normal on the Screening laboratory assessments, or other clinically significant laboratory abnormalities, which in the opinion of the Investigator may prevent the subject from safely participating in study.
12. Participants with a history of risk factors of Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) or an ECG demonstrating a Fridericia's corrected QT interval (QTcF) >450 msec in males and QTcF > 470 in females at screening.
13. Significant symptoms, medical conditions, or other circumstances which, in the opinion of the Investigator, would preclude compliance with the protocol, adequate cooperation in the study or obtaining informed consent, or may prevent the subject from safely participating in study. This includes, but is not limited to, subjects with attention deficit hyperactivity disorder receiving central stimulants (e.g. methylphenidate or other central stimulants), as well as subjects with severe respiratory insufficiency, respiratory depression, airway obstruction, gastrointestinal motility disorders, severe hepatic insufficiency, planned surgery and prior treatment with monoamine oxidase inhibitors.
14. Is an employee of the Investigator or the trial site, with direct involvement in the proposed trial or other studies under the direction of the Investigator or trial site, or is a family member of an employee or of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2015-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frost, MD, Principal Investigator — Frost Medical Group
Locations (32):
- United States (10):
  - Parkway Medical Center, Birmingham, Alabama
  - Haleyville Clinical Research LLC, Haleyville, Alabama
  - Boyett Health Services Inc, Hamilton, Alabama
  - Dr Vijapura and Associates, Jacksonville, Florida
  - TRY Research, Maitland, Florida
  - Stanley Street Treatment and Resources Inc, Fall River, Massachusetts
  - Wellness and Research Center, Belvidere, New Jersey
  - Comprehensive Clinical Research, Berlin, New Jersey
  - STARS/Columbia University, New York, New York
  - Frost Medical Group, LLC, Conshohocken, Pennsylvania
- Australia (4):
  - Newcastle Community Health Services, Newcastle
  - Drug & Alcohol Services SA Drug and Alcohol Services, Norwood
  - Royal Prince Alfred Hospital, Sydney
  - South Eastern Sydney Local Health District (SESLHD), Sydney
- Denmark (2):
  - Center for Misbrugsbehandling, Aarhus
  - Behandlingscenter Odense, Odense
- Germany (5):
  - Gemeinschaftspraxis Schnaitmann/Schaffert Salzstrasse, Heilbronn
  - Studikum - Zentrum fur Klinische Studien im Praxiszentrum Friedrichsplatz, Kassel
  - Klinik fur Abhangiges Verhalten und Suchtmedizin Zentralinstitut, Mannheim
  - Psychosoziale Begleitung - Praxis Boniakowski, Regensburg
  - Praxisgemeinschaft, Stuttgart
- Hungary (2):
  - Clinexpert Kft, Budapest
  - XVI. Kerület Kertvárosi Egészségügyi Szolgálata, Addiktológia, Budapest
- Sweden (2):
  - Metadonsektionen, Stockholm
  - Centrallasarettet Vasteras, Västerås
- Taiwan (3):
  - Jinan Psychiatric Center, Ministry of Health and Welfa, Tainan, Tainan County
  - China Medical University Hospita, Taichung
  - Taipei City Hospital, Taipei
- United Kingdom (4):
  - Blackberry Centre Blackberry Hill Hospital, Fishponds, Bristol
  - Hellesdon Hospital The Weavers Centre, Hellesdon, Norwich
  - NHS Tayside, Dundee
  - Lambeth Drug and Alcohol Service Lorraine Hewitt House, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frost M, Bailey GL, Lintzeris N, Strang J, Dunlop A, Nunes EV, Jansen JB, Frey LC, Weber B, Haber P, Oosman S, Kim S, Tiberg F. Long-term safety of a weekly and monthly subcutaneous buprenorphine depot (CAM2038) in the treatment of adult out-patients with opioid use disorder. Addiction. 2019 Aug;114(8):1416-1426. doi: 10.1111/add.14636. Epub 2019 Jun 3. PMID 31013390

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient enrolled in the study but did not receive CAM2038
Groups:
- CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX: Subjects previously exposed to SL BPN/NX who received CAM2038 q1w or q4w
- CAM2038 q1w or q4w New to BPN Treatment: New to BPN Treatment who received CAM2038 q1w or q4w
Period: Overall Study
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Started | 190 | 37
Completed Treatment | 138 | 29
Completed | 132 | 25
Not Completed | 58 | 12

BASELINE CHARACTERISTICS:
Groups:
- CAM2038 q1w or q4w New to BPN Treatment: New to BPN Treatment who received CAM2028 q1w or q4w
- Total: Total of all reporting groups
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment | Total
Number analyzed (Participants) | 190 | 37 | 227
Age, Continuous [Mean (Full Range); unit: years] | 41.3 [24 to 66] | 41.8 [24 to 61] | 41.4 [24 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 13 | 84
  Male | 119 | 24 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 187 | 35 | 222
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 17 | 20
  White | 183 | 20 | 203
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 36 | 127
  Europe | 76 | 0 | 76
  Australia | 23 | 1 | 24
BMI (kg/m^2) [Mean (Full Range); unit: kg/m^2] | 26.7 [16.9 to 50.4] | 25.3 [18.2 to 46.4] | 26.5 [16.9 to 50.4]

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Treatment-Emergent Adverse Events (TEAE) During the Treatment Period-Overall Safety Population
Description: Subjects With Treatment-Emergent Adverse Events (TEAE) During the Treatment Period. Safety Assessments: Adverse events (AEs) and serious adverse events (SAEs)-Overall Safety Population
Time Frame: 12 months- 48 week
Population: Overall Safety Population-Subjects treated with CAM2038
Measure: Number; unit: participants
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Number analyzed (Participants) | 190 | 37
participants
  Subject had at least 1 TEAE | 131 | 12
  Subject had at least 1 drug-related TEAE | 58 | 2
  Subject had at least 1 severe TEAE | 13 | 2
  Deaths | 0 | 0
  Subject had at least 1 non-fatal SAE | 10 | 2
  Subject had at least 1 non-fatal drug related SAE | 0 | 0
  Hospitalizations | 9 | 1
  Subject discontinued study drug due to a TEAE | 4 | 1

2. Primary Outcome: Subjects With Treatment-Emergent Adverse Events (TEAE) During the Treatment Period-Full Exposure Safety Population
Description: Subjects With Treatment-Emergent Adverse Events (TEAE) During the Treatment Period. Safety Assessments: Adverse events (AEs) and serious adverse events (SAEs)-Full Exposure Safety Population
Time Frame: 12 months- 48 week
Population: Full Exposure Safety Population-Subjects treated with CAM2038
Measure: Number; unit: participants
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Number analyzed (Participants) | 128 | 28
participants
  Subject had at least 1 TEAE | 95 | 8
  Subject had at least 1 drug-related TEAE | 41 | 1
  Subject had at least 1 severe TEAE | 11 | 1
  Deaths | 0 | 0
  Subject had at least 1 non-fatal SAE | 8 | 1
  Subject had at least 1 non-fatal drug related SAE | 0 | 0
  Hospitalizations | 7 | 1
  Subject discontinued study drug due to a TEAE | 0 | 0

3. Secondary Outcome: Mean Percentage of Negative Urine Toxicology Results for Illicit Opioid Use Supported by Self Reported Illicit Opioid Use (Efficacy Population)
Description: The following is a summary of Mean Percentage of Negative Urine Toxicology Results for Illicit Opioid Use Supported by Self Reported Illicit Opioid Use (Efficacy Population)
Time Frame: 12 months (48 weeks)
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: percentage of negative urine samples
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Number analyzed (Participants) | 189 | 37
percentage of negative urine samples | 82.8 (29.31) | 41.2 (34.04)

4. Secondary Outcome: Mean Percentage of Self-reported No Illicit Opioid Use (Efficacy Population)
Description: The following is a summary of Mean Percentage of Self-Reported No Illicit Opioid Use during the entire study (Efficacy Population). The proportion of patients who reported no illicit opioid use during the study was analyzed. For example if a subject provided 10 self reports and 2 out of the 10 were "Used", the percentage for the subject would be 20%. The average percentage of all patients is provided.
Time Frame: 12 months (48 weeks)
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: Mean percentage of no illicit opioid use
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Number analyzed (Participants) | 188 | 37
Mean percentage of no illicit opioid use | 92.5 (19.78) | 74.0 (31.28)

5. Secondary Outcome: Summary of Retention in Treatment (Efficacy Population)
Description: The following is a summary of treatment retention over 48 weeks
Time Frame: 48 weeks of treatment
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Number analyzed (Participants) | 190 | 37
weeks | 38.3 (16.85) | 43.6 (11.50)

6. Secondary Outcome: Summary of Clinical Opiate Withdrawal Scale (COWS) at Selected Time Points (Efficacy Population)
Description: A summary of COWS (administered by the Clinician) over 48 weeks to show withdrawal symptoms from baseline to end of treatment. This scale consists of 11 common opiate withdrawal signs or symptoms, rated on a numeric scale from 0 to 4 or 5 and based on a timed period of observation of the subject by the rater. Higher scores are associated with greater withdrawal symptoms with a total range for all items of between 0-48
Time Frame: 12 months- 48 week
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Number analyzed (Participants) | 190 | 37
score on a scale
  Baseline | 2.0 (2.7) | 10.6 (3.7)
  Visit 3 Day 8: number analyzed (Participants) | 103 | 36
  Visit 3 Day 8 | 3.7 (4.1) | 3.0 (2.5)
  Visit 26 Day 169: number analyzed (Participants) | 114 | 26
  Visit 26 Day 169 | 1.9 (2.8) | 0.2 (0.4)
  End of Treatment | 1.4 (2.3) | 0.3 (0.5)

7. Secondary Outcome: Summary of Subjective Opiate Withdrawal Scale (SOWS) at Selected Time Points (Efficacy Population)
Description: Summary of SOWS over time to show withdrawal symtons, from baseline to end of treatment. This form contains 16 questions that rate the intensity of withdrawal from 0 ("Not at all") to 4 ("Extremely"), with higher scores associated with greater withdrawal symptoms and total range for all items of 0-64
Time Frame: 12 months- 48 week
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Number analyzed (Participants) | 190 | 37
score on a scale
  Baseline | 4.7 (8.1) | 27.1 (15.3)
  Visit 3 Day 8: number analyzed (Participants) | 103 | 36
  Visit 3 Day 8 | 8.4 (11.5) | 8.9 (10.9)
  Visit 26 Day 169: number analyzed (Participants) | 114 | 26
  Visit 26 Day 169 | 4.3 (7.2) | 3.0 (7.5)
  End of Treatment: number analyzed (Participants) | 138 | 29
  End of Treatment | 3.3 (6.3) | 3.9 (8.0)

8. Secondary Outcome: Summary of Desire to Use Visual Analog Scale (VAS) at Selected Time Points (Efficacy Population)
Description: The following table summarizes the desire to use measurements over a period of 12 months - 48 weeks. Desire to Use assessments were administered using a unipolar 100 mm VAS. Subjects were asked "Since your last scheduled assessment visit, indicate your worst or strongest desire to use opioids, where 0 = No desire to use and 100 mm = Strongest possible desire.
Time Frame: 12 months- 48 week
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Number analyzed (Participants) | 190 | 37
score on a scale
  Baseline: number analyzed (Participants) | 189 | 37
  Baseline | 11.7 (24.2) | 74.8 (24.8)
  Visit 3 Day 8: number analyzed (Participants) | 103 | 36
  Visit 3 Day 8 | 18.8 (29.8) | 23.0 (25.9)
  Visit 26 Day 169: number analyzed (Participants) | 113 | 26
  Visit 26 Day 169 | 6.4 (15.6) | 5.8 (16.7)
  End of Treatment: number analyzed (Participants) | 138 | 28
  End of Treatment | 6.4 (16.5) | 2.8 (6.2)

9. Secondary Outcome: Summary of Need to Use Visual Analog Scale (VAS) at Selected Time Points (Efficacy Population)
Description: The following results summarize the need to use VAS over a period of 12 months - 48 weeks. Need to Use assessments were administered using a unipolar 100 mm VAS. Subjects were asked "Since your last scheduled assessment visit, indicate your worst or strongest need to use opioids, where 0 = No need to use and 100 mm = Strongest possible need.
Time Frame: 12 months- 48 week
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
Number analyzed (Participants) | 190 | 37
score on a scale
  Baseline | 11.7 (23.8) | 76.3 (24.9)
  Visit 3 Day 8: number analyzed (Participants) | 103 | 36
  Visit 3 Day 8 | 18.0 (27.9) | 34.3 (29.2)
  Visit 26 Day 169: number analyzed (Participants) | 114 | 26
  Visit 26 Day 169 | 5.6 (12.5) | 8.0 (18.2)
  End of Treatment: number analyzed (Participants) | 138 | 28
  End of Treatment | 5.4 (14.3) | 5.3 (15.9)

ADVERSE EVENTS:
Time Frame: Time frame of adverse events was 12 months - 48 weeks.
Groups:
- CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX: Subjects exposed to SL BPN/NX who received CAM2038 q1w or q4w
- CAM2038 q1w or q4w New to BPN Treatment: New to BPN Treatment who received either CAM2028 q1w or q4w
Arm/Group | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX | CAM2038 q1w or q4w New to BPN Treatment
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/37
Serious Adverse Events (participants affected / at risk) | 13/190 | 2/37
Other Adverse Events (participants affected / at risk) | 131/190 | 11/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX (N=190) | CAM2038 q1w or q4w New to BPN Treatment (N=37)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM2038 q1w or q4w With Prior Exposure to SL BPN/NX (N=190) | CAM2038 q1w or q4w New to BPN Treatment (N=37)
Injection site Pain (General disorders) | 33 (33) | 2 (2)
Injection SIte Swelling (General disorders) | 25 (25) | 2 (2)
Injection site erythema (General disorders) | 20 (20) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (16) | 0 (0)
Headache (Nervous system disorders) | 18 (18) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (12) | 0 (0)
Nasopharyngitis (Infections and infestations) | 17 (17) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (9) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT02672111/SAP_000.pdf
  • Study Protocol (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT02672111/Prot_001.pdf